CLINICAL TRIAL: NCT01281722
Title: Role of SLURP-1 in Melanoma and Melanoma Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shiou-Hwa Jee, M.D., Ph.D., Professor,Department of Dermatology,National Taiwan University Hospital
Other Study IDs: 201012044RB
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Melanoma;
Keywords: healthy adults; melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, DNA, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy adults: healthy adults with the age among 20 to 95 years old
- melanoma cases: the people who are diagnosed melanoma in NTU hospital

SUMMARY:
Melanoma is the most aggressive skin cancer, with a propensity to metastasize, and is resistant to most of the current therapeutic regimens. Incidence rate of melanoma in patients with MDM (Mal De Maleda, with SLURP-1 mutation) is much higher than normal counterpart. SLURP-1 (lymphocyte antigen 6/urokinase-type plasminogen activator receptor related protein-1) is an allosteric agonist to the nicotinic acetylcholine receptor (nAchR) and it regulates epidermal homeostasis and T-cell function. The preliminary results of comparing human peripheral blood mononuclear cells (PBMCs) from 4 affected and 15 unaffected members from the family with MDM revealed that T-cell activation was impaired in PBMCs with the heterozygous and homozygous SLURP-1 G86R mutation. (2 of affected members developed melanoma.) Since there is currently no effective treatment for metastatic melanoma, identifying novel molecular mechanisms may lead to development of new treatments for metastatic melanomas.

Previous study showed that melanoma stem cells (MSCs) are crucial in melanoma pathogenesis: 1.Melanoma contains ABCB5, CD133 and ABCG2 positive cells had enhanced tumorigenic potential. 2.Higher frequencies of cells capable of initiating melanoma xenografts when using IL2Rγ-/- NOD SCID mice. These data confirmed the interaction between T cells and MSCs.

In this project, we will investigate the roles of SLURP-1 in melanoma and MSCs. Investigating and verifying the interaction between T-cells from patients with MDM and melanoma cells to confirm the SLURP-1 function of tumorigenesis in xenotransplant mice (IL2Rγ-/- NOD SCID) model. To reveal the role of SLURP-1 silencing in melanoma cell lines by using not only A2058 , A375 and MeWo mwlanima cell lines but also ABCB5+ melanoma cells and ABCB5- melanoma cells through the tumorigenesis, apoptosis,angiogenesis, proliferation, melanosphere formation assays.

The aim of this project is to investigate the roles and molecular mechanisms of SLURP-1 in melanoma carcinogenesis, which may improve the development of novel treatments for melanoma.

DETAILED DESCRIPTION:
Cutaneous melanoma is an aggressive neoplasm refractory to traditional therapies, especially at the metastatic stage. Furthermore, its incidence is continuously increasing during the last decade (1). Melanomas develop through a multistep process that from normal melanocytes proceeds to nevi and to radial and vertical growth phase tumors (2). During this process, melanomas are characterized by certain well-defined genetic alterations as well as frequent chromosomal aberrations associated with tumor progression (3). However, the molecular mechanisms involved in the carcinogenesis and progression of melanoma are complex and not entirely clear (4). Because of the intractability of metastatic melanomas with only 14% of the patients survive for 5 years and no effective treatments (2), understanding the underlying molecular mechanisms involved in melanoma and identifying molecular markers may lead to improvements in therapeutic approaches for metastatic melanomas.

Mal de Meleda (MDM; OMIM 248300) is a rare autosomal recessive disorder characterized by erythema and hyperkeratosis of the palms and soles, extending to the dorsal aspects of the hands and feet (known as transgrediens), and perioral erythema and psoriasiform plaques on the elbows and knees. (5-7) Homozygous mutations of the SLURP1 gene (previously known as ARS component B) encoding lymphocyte antigen 6/urokinase-type plasminogen activator receptor related protein-1 (SLURP-1) have been identified as the cause of MDM. (8-10) Mutations of the SLURP1 gene affect the expression, integrity and stability of SLURP-1 on the upper layer of the epidermis and in cultured mature keratinocytes. (11) Other studies also demonstrated that SLURP-1 acts as a positive allosteric ligand for 7-nAchR in keratinocytes, eliciting proapoptotic activity and differentiation. (12,13) As well as in epidermis and keratinocytes, the expression of SLURP-1 has been found in T cells, B cells, dendritic cells and macrophages. (14-15) Malignant melanoma (MM) has been reported to be the predominant cutaneous malignancy occurring in the hyperkeratotic area in patients with MDM. (16) The incidence of MM in MDM is significantly higher than in the general population.(17) At least six cases of MM have been reported in patients with MDM;27-29 two of the reported cases were siblings. (18) The possible explanations of the higher incidence of MM in patients with MDM include: (i) lack of proapoptotic effect of SLURP-1; (ii) defective T-cell activation and tumour monitoring; or (iii) prolonged inflammation in hyperkeratotic skin.

The previous study showed that peripheral blood mononuclear cells (PBMCs) with the heterozygous and homozygous SLURP-1 G86R mutation had defective T-cell activation. This was restored by the addition of 0•5 μg mL-1 recombinant human SLURP-1 protein. (19) Previous study showed that a putative monoclonal antibody that recognized ABCB5 was used to isolate melanoma stem cells (MSCs). (20) In this study, the investigators will investigate the roles of SLURP-1 in melanoma cells (including MSC) and also its interaction between melanoma cells and T-cells.

Aims：

1. To evaluate the significance and correlation of SLURP-1 expression in melanoma cells and melanoma metastasis in human tissues and mouse metastasis models.
2. To assess the function of the SLURP-1 protein in melanoma cells and melanoma stem cells.
3. To investigate the interaction between T-cells with SLURP-1 mutation and melanoma cells / MSCs.
4. Confirm the biological effects of SLURP-1 on melanoma cells / MSCs.
5. To investigate the relationship between SLURP-1 overexpression and melanoma cancer biology.

References

1. Gray-Schopfer V, Wellbrock C, Marais R. Melanoma biology and new target therapy. Nature 2007; 445: 851-7.
2. Miller AJ, Mihm MC. Melanoma. N Engl J Med 2006; 355: 51-65.
3. Jonsson G, et al. Genomic profiling of malignant melanoma using tiling-resolution array CGH. Oncogene 2007; 6: 4738-48.
4. Bemis LT, Chen R, Amato CM et al. MicroRNA-137 targets microphthalmia-associated transcription factor in melanoma cell lines. Cancer Res 2008; 68: 1362-8.
5. Lucker GP, Van De Kerkhof PC, Steijlen PM. The hereditary palmoplantar keratoses: an updated review and classification. Br J Dermatol 1994; 131:1-14.
6. Bergman R, Bitterman-Deutsch O, Fartasch M et al. Mal de Meleda keratoderma with pseudoainhum. Br J Dermatol 1993; 128:207-12.
7. Jee SH, Lee YY, Wu YC et al. Report of a family with mal de Meleda in Taiwan: a clinical, histopathological and immunological study. Dermatologica 1985; 171:30-7.
8. Fischer J, Bouadjar B, Heilig R et al. Mutations in the gene encoding SLURP-1 in Mal de Meleda. Hum Mol Genet 2001; 10:875-80.
9. Ward KM, Yerebakan O, Yilmaz E et al. Identification of recurrent mutations in the ARS (component B) gene encoding SLURP-1 in two families with mal de Meleda. J Invest Dermatol 2003; 120:96-8.
10. Mastrangeli R, Donini S, Kelton CA et al. ARS component B: structural characterization, tissue expression and regulation of the gene and protein (SLURP-1) associated with mal de Meleda. Eur J Dermatol 2003; 13:560-70.
11. Favre B, Plantard L, Aeschbach L et al. SLURP1 is a late marker of epidermal differentiation and is absent in mal de Meleda. J Invest Dermatol 2007; 127:301-8.
12. Grando SA. Basic and clinical aspects of non-neuronal acetylcholine: biological and clinical significance of non-canonical ligands of epithelial nicotinic acetylcholine receptors. J Pharmacol Sci 2008; 106:174-9.
13. Arredondo J, Chernyavsky AI, Webber RJ et al. Biological effects of SLURP-1 on human keratinocytes. J Invest Dermatol 2005; 125:1236-41.
14. Moriwaki Y, Yoshikawa K, Fukuda H et al. Immune system expression of SLURP-1 and SLURP-2, two endogenous nicotinic acetylcholine receptor ligands. Life Sci 2007; 80:2365-8.
15. Kawashima K, Yoshikawa K, Fujii YX et al. Expression and function of genes encoding cholinergic components in murine immune cells. Life Sci 2007; 80:2314-19.
16. Nakajima K, Nakano H, Takiyoshi N et al. Papillon-Lefèvre syndrome and malignant melanoma. A high incidence of melanoma development in Japanese palmoplantar keratoderma patients. Dermatology 2008; 217:58-62.
17. Sartore L, Bordignon M, Bassetto F et al. Melanoma in skin affected with keratoderma palmoplantaris hereditaria (mal de Meleda): treatment with excision and grafting. J Am Acad Dermatol 2009; 61:161-3.
18. Mozzillo N, Nunziata CA, Caraco C et al. Malignant melanoma developing in an area of hereditary palmoplantar keratoderma (mal de Meleda). J Surg Oncol 2003; 84:229-33.
19. Tjiu JW, Lin PJ, Wu WH et al. SLURP1 mutation-impaired T-cell activation in a family with mal de Meleda. Br J Dermatol. 2010 Sep 21
20. Schatton T, Murphy GF, Frank NY et al. Identification of cells initiating human melanomas. Nature. 2008 Jan 17;451(7176):345-9

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of melanoma Disease by NTU hospital(group of cases)
* healthy adults(groups of control)

Exclusion Criteria:

* two groups whose age are younger than 20 or older tha 95 years old
* Clinical diagnosis of non-melanoma Disease by NTU hospital(group of cases)

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: case and control study of melanoma disease
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-07 (Estimated); Study Completion 2019-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shiou-Hwa Jee, M.D., Ph.D., Study Chair — Department of Dermatology, National Taiwan University Hospital.
Locations (1):
- Department of Dermatology, National Taiwan University Hospital., Taipei, Taiwan